CLINICAL TRIAL: NCT03231488
Title: The Effect of Mindfulness on Stimulus Over-selectivity and Selective Attention to Threat Following Acquired Brain Injury
Brief Title: The Effect of Mindfulness on Cognition and Emotion Following Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Cambridgeshire Community Services NHS Trust (Other); Cambridgeshire and Peterborough NHS Foundation Trust (Other); NORFOLK COMMUNITY HEALTH AND CARE NHS TRUST (Unknown); Northamptonshire Healthcare NHS Foundation Trust (Other); Headway Cambridgeshire (Unknown); Headway Essex (Unknown); Headway Norfolk and Waveney (Unknown); Icanho, Livability (Unknown); Brain Injury Rehabilitation Trust (Other); St Andrew's Healthcare (Other); Partnerships in Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS project ID: 213205
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-06

CONDITIONS: Injuries, Brain
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness intervention (Experimental)
  Interventions: Other: Mindfulness intervention
- Control intervention (unfocused attention) (Active Comparator)
  Interventions: Other: Control intervention (unfocused attention)

INTERVENTIONS:
Other: Mindfulness intervention — A 10 minute mindfulness of breath exercise
  Arms: Mindfulness intervention
Other: Control intervention (unfocused attention) — A 10 minute unfocused attention intervention - participants are asked to let their mind wander on anything that comes to mind.
  Arms: Control intervention (unfocused attention)

SUMMARY:
Can mindfulness help with attention and emotion difficulties after a brain injury?

People who have a brain injury often have problems with their attention and emotions. This study will see if a short mindfulness task can help with these problems. So far, there are not many studies looking at this and those that do show mixed results. When being mindful someone is aware of their attention and focuses on the present moment without passing judgement. This study focuses on over-selectivity and selective attention to threat after a brain injury. These are two concepts involved in attention and emotion problems. Over-selectivity is when someone focuses on only one thing around them and misses other key things. Selective attention to threat is when someone's focus is drawn to something around them that is seen as threatening. This has been shown to cause and keep anxious feelings going. This research will see if a short mindfulness task can help those with a brain injury by reducing overselectivity and selective attention to threat on two tasks. Participants will be recruited from NHS and non-NHS brain injury services. The study will take around two hours to complete for each participant. In summary, this study looks to see if a specific mindfulness exercise can be helpful for specific attention and emotion problems. It could be a first step in making treatment better and giving more treatment options for those with a brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Medical evidence of ABI with attention or executive functioning difficulties, such as difficulties with planning, inhibition or attention
* Time since ABI to be 9 months or greater • ABI severity to be moderate to severe, determined by the Mayo classification system (Malec et al., 2007). This is classification system is frequently used to determine ABI severity and is standard practice to record at the acute stage of care when the individual is admitted to hospital. This means there must be evidence of one or more of the following in medical notes: the individual's lowest Glasgow Coma Scale (GCS) score is less than 13, there is a loss of consciousness of at least 30 minutes immediately following ABI and post traumatic amnesia (PTA) is at least 24 hours in length. If there is no evidence of this in the medical notes, then there must be evidence that the individual has clinically significant difficulties resulting from their ABI to have needed a referral to brain injury services.
* There are self-reported or clinician-identified emotional difficulties to adjusting to circumstances post-ABI

Exclusion Criteria:

* Significant, severe and enduring presence of mental health difficulties or substance misuse that would prevent valid engagement in experimental tasks
* Perceptual, language, communication, reading or motor difficulties that would prevent valid engagement in experimental tasks
* The presence of developmental or acquired dyslexia affecting the automatic reading of words in the emotional Stroop
* Severe cognitive difficulties that would prevent valid engagement in experimental tasks
* Presence of pre-existing or comorbid disorders that may affect cognitive functioning (other than ABI) that would prevent valid engagement in experimental tasks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Emotional Stroop | Administered pre- and post- 10-minute intervention, so over a period of one hour
  This will be a computer task that measures selective attention to threat.
  In the emotional Stroop, different coloured words are presented to participants and the emotional meaning of the words are manipulated. Participants are instructed to name the colour of the words as quickly as possible, whilst ignoring the meaning of the words. Selective attention to threat will be inferred when word colour-naming takes longer when the meaning of the word is threatening relative to neutral. So, the greater the difference between reaction times to neutral and threatening words, the greater the selective attention to threat.
Over-selectivity task. | Administered pre- and post- 10-minute intervention, so over a period of one hour
  This will be a computer task that measures over-selectivity.
  Practice phase - two cards, each with two images appear on the screen. One card is the correct one to select and the other is incorrect. This happens for two sets of two cards (pair 1 and pair 2). Test phase - participants are presented with two single stimuli simultaneously, one from the reinforced compound and one from the verbally punished compound (Figure 4). They are instructed to select one of the pictures on the screen.
  Over-selectivity will occur if participants fail to learn about one of the stimuli in the previously reinforced compound and therefore fail to select that stimuli they had not learned about in the practice phase.
  So, the higher the score on the over-selectivity task, the greater the difference between the most and least chosen stimuli, which means that the participant is demonstrating greater over-selectivity.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Pre-intervention (baseline measure)
  A self-report measure consisting of 14 items. The measure gives an overall score, as well as separate scores for severity of anxiety and depression subscales.
The Five Facet Mindfulness Questionnaire (FFMQ) | Pre-intervention (baseline measure)
  This will be used to characterise levels of mindfulness. This is a self-report measure, consisting of 39 items.
Test of Everyday Attention (TEA) | Pre-intervention (baseline measure)
  Subtests will be used to measure baseline measures of attention. Elevator counting is a measure of sustained attention and elevator counting with distraction is a measure of selective attention.
Weschler Test of Adult Reading (WTAR) | Pre-intervention (baseline measure)
  This will be used to measure a baseline measure of pre-morbid functioning. Participants read a list of 50 words with irregular pronunciations to assess previous learning of the words.

CONTACTS AND LOCATIONS:
Locations (12):
- United Kingdom (12):
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Cambridgeshire Community Services Nhs Trust, Cambridge
  - Headway Cambridgeshire, Cambridge
  - Brain Injury Rehabilitation Trust, Ely
  - Headway Essex, Essex
  - Headway Norfolk & Waveney, Norfolk
  - Norfolk Community Health and Care Nhs Trust, Norfolk
  - Northamptonshire Healthcare Nhs Foundation Trust, Northampton
  - Partnerships in Care, Northampton
  - St Andrews Healthcare, Northampton
  - Cambridgeshire and Peterborough Nhs Foundation Trust, Peterborough
  - Icanho, Livability, Stowmarket